CLINICAL TRIAL: NCT06901102
Title: Bee Venom As Immunomodulator and Its Effect on Chronic Kidney Disease-Mineral Bone Disorders in Hemodialysis Patients: a Prospective Randomized Controlled Trial
Brief Title: Effect of Bee Venom on Chronic Kidney Disease-Mineral Bone Disorders in Hemodialysis Patients: a Randomized Controlled Trial
Acronym: BeeVenom-CKD
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Islam Mohammed Ahmed Aboalela, Nephrology Resident, Urology and Nephrology Center, Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS.24.12.3035
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Disease; Bee Venom; Hemodialysis
Keywords: Bee venom; Mineral bone disorder; Hemodialysis; Immunomodulation; Regulatory T cells; Bone turnover markers
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Bee Venoms; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bee Venom Injection (Intervention Group) (Experimental): This group will receive bee venom injections to evaluate its effect on chronic kidney disease-related mineral bone disorder in hemodialysis patients. The bee venom will be administered subcutaneously, starting with a dose of 0.05 mL three times a week and escalating to 0.5 mL by week 5. The treatment will last for six months.
  Interventions: Drug: Bee Venom Injection
- Standard Care (Control Group) (Active Comparator): This group will receive the usual clinical care for mineral bone disorders associated with chronic kidney disease in hemodialysis patients. Standard care may include phosphate binders, vitamin D receptor activators, and other treatments commonly used to manage MBD in CKD patients.
  Interventions: Drug: Standard Care for CKD-MBD

INTERVENTIONS:
Drug: Bee Venom Injection — This intervention involves the administration of purified bee venom from Apis mellifera species (Abevac) via subcutaneous injections. The dosage starts at 0.05 mL three times a week and gradually escalates to 0.5 mL three times a week by week 5. The total duration of the treatment is 6 months. Bee venom is being evaluated for its potential immunomodulatory effects, including enhancing regulatory T cell function and improving mineral bone disorder (MBD) in patients undergoing hemodialysis.
  Arms: Bee Venom Injection (Intervention Group)
Drug: Standard Care for CKD-MBD — This intervention represents the standard care for patients with chronic kidney disease-mineral bone disorder (CKD-MBD) undergoing hemodialysis. The treatment typically includes phosphate binders to control phosphorus levels, vitamin D receptor activators to regulate calcium and phosphorus metabolism, and calcimimetics to control parathyroid hormone (PTH) levels. The specific regimen may vary according to individual patient needs, but the control group will not receive bee venom injections as part of their therapy.
  Arms: Standard Care (Control Group)

SUMMARY:
This study aims to evaluate the effectiveness of bee venom injections as a treatment for chronic kidney disease (CKD)-mineral bone disorder (MBD) in patients undergoing hemodialysis. MBD is a common complication in CKD patients, leading to abnormal mineral metabolism, bone disease, and increased cardiovascular risks. Current treatments are often inadequate and can have significant side effects.

In this study, we will compare the effects of bee venom injections with standard care treatments in hemodialysis patients. Bee venom is known for its potential anti-inflammatory and immunomodulatory properties, which may help improve mineral metabolism and bone health regulation in these patients. By stimulating regulatory T cells (Tregs) through bee venom, we aim to reduce inflammation and restore bone health.

We hope to answer whether bee venom can effectively reduce mineral bone disorder markers (such as calcium, phosphorus, and parathyroid hormone levels) and improve bone density in hemodialysis patients. The results could lead to a new treatment option for CKD-MBD, improving patient outcomes and quality of life.

DETAILED DESCRIPTION:
This prospective, randomized controlled trial investigates the potential therapeutic role of bee venom in improving mineral bone disorder (MBD) among hemodialysis patients with chronic kidney disease (CKD). MBD is a common complication in CKD, characterized by disruptions in calcium, phosphorus, parathyroid hormone (PTH), and vitamin D metabolism, leading to abnormal bone remodeling and an increased risk of fractures and cardiovascular events. Conventional treatments for MBD, including phosphate binders, vitamin D analogs, and calcimimetics, often fall short in achieving optimal biochemical control and carry significant side effects. Therefore, there is a need for innovative therapies.

Bee venom, derived from the sting of the honeybee (Apis mellifera), has shown immunomodulatory and anti-inflammatory properties, which may play a role in modulating immune responses and regulating mineral metabolism. Previous studies suggest that bee venom can influence T cell activity, particularly enhancing the function of regulatory T cells (Tregs), which are known to suppress inflammation and help maintain immune balance. Given that inflammation is a key driver in the pathogenesis of MBD, targeting the immune system through bee venom presents a novel approach to improving bone and mineral metabolism.

The study will involve 60 patients undergoing maintenance hemodialysis, randomly assigned to either the intervention group receiving bee venom injections or the control group receiving standard care. Bee venom will be administered subcutaneously, with a dose escalation schedule starting at 0.05 mL three times weekly in the first week and increasing to 0.5 mL three times weekly by week 5. The treatment will last for six months.

Clinical and laboratory evaluations will assess the effects of bee venom on key MBD biomarkers, including serum calcium, phosphorus, PTH levels, and bone turnover markers. Radiological assessments using quantitative computed tomography (QCT) will evaluate bone mineral density changes at the lumbar vertebrae. The study will also assess the safety profile of bee venom by monitoring adverse events and allergic reactions.

The primary goal is determining whether bee venom can significantly improve MBD markers compared to standard care. Secondary objectives include evaluating changes in bone mineral density, assessing the safety and tolerability of bee venom, and exploring potential effects on inflammation markers and cardiovascular risk factors. The findings from this study may provide insights into the possible role of bee venom as a therapeutic agent in managing CKD-MBD. They could lead to a new treatment option for hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged 18 years and older.
* Patients undergoing maintenance hemodialysis three times weekly for at least six months.
* Patients who are not scheduled for kidney transplantation within the next year.

Exclusion Criteria:

* Current pregnancy or lactation.
* Medical history of chronic conditions such as liver disease, cancer, or autoimmune diseases.
* Refusal to participate in the study.
* Active chronic infections, including HIV, HCV, HBV, and tuberculosis.
* Current use of medications affecting bone metabolism (e.g., calcitonin, denosumab, estrogen) within the last six months.
* History of renal allograft failure within the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Improvement in Bone-Specific Biomarkers (BALP, P1NP, TRAP-5b) | 6 months The primary outcome will be assessed at baseline and after 6 months of treatment to evaluate the effect of bee venom on bone metabolism in CKD-MBD patients undergoing hemodialysis.
  The primary outcome measure will evaluate the effect of bee venom injections on bone-specific biomarkers in hemodialysis patients with chronic kidney disease-mineral bone disorder (CKD-MBD). This will be assessed by measuring changes in bone-specific alkaline phosphatase (BALP), propeptides of type I procollagen (P1NP), and tartrate-resistant acid phosphatase (TRAP-5b) levels from baseline to the end of the study. The aim is to determine if bee venom therapy can improve bone turnover markers compared to standard care.

SECONDARY OUTCOMES:
Change in Bone Mineral Density (BMD) Measured by QCT of Lumbar Vertebrae | 6 months Bone mineral density measurements will be taken at baseline and at the end of the 6-month treatment period to assess the impact of bee venom on bone health in CKD-MBD patients undergoing hemodialysis.
  The secondary outcome measure will evaluate the effect of bee venom injections on bone mineral density (BMD) in hemodialysis patients with CKD-MBD, measured by quantitative computed tomography (QCT) of the lumbar vertebrae. Changes in both cortical and trabecular bone density will be assessed from baseline to the end of the study. This will help determine if bee venom therapy has a beneficial effect on improving bone density compared to standard care.

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Mansoura University, Al Mansurah, Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
At this stage, we have not yet determined whether individual participant data (IPD) will be shared with other researchers. After the study is completed, we will assess the feasibility and ethical considerations regarding data sharing. If IPD sharing becomes an option, appropriate measures will be taken to ensure participant confidentiality and compliance with data protection regulations.

REFERENCES:
- [Background] Waziri B, Duarte R, Naicker S. Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD): Current Perspectives. Int J Nephrol Renovasc Dis. 2019 Dec 24;12:263-276. doi: 10.2147/IJNRD.S191156. eCollection 2019. PMID 31920363
- [Background] An HJ, Kim JY, Kim WH, Han SM, Park KK. The Protective Effect of Melittin on Renal Fibrosis in an Animal Model of Unilateral Ureteral Obstruction. Molecules. 2016 Aug 27;21(9):1137. doi: 10.3390/molecules21091137. PMID 27618890
- [Background] Hwang DS, Kim SK, Bae H. Therapeutic Effects of Bee Venom on Immunological and Neurological Diseases. Toxins (Basel). 2015 Jun 29;7(7):2413-21. doi: 10.3390/toxins7072413. PMID 26131770
- [Background] Carpena M, Nunez-Estevez B, Soria-Lopez A, Simal-Gandara J. Bee Venom: An Updating Review of Its Bioactive Molecules and Its Health Applications. Nutrients. 2020 Oct 31;12(11):3360. doi: 10.3390/nu12113360. PMID 33142794